CLINICAL TRIAL: NCT01105156
Title: Outcomes of Gastric Band Fills as Found With a Patient Self-reported Questionnaire. The VEW [Vomiting, Eating, and Weight Loss] Questionnaire
Brief Title: Outcomes of Gastric Band Fills as Found With a Patient Self-reported Questionnaire: The Vomiting, Eating, and Weight Loss (VEW) Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: North Eastern Weight Loss Surgery (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Patrick Moore, North Eastern Weight Loss Surgery
Other Study IDs: NEWLS29401
Record Dates: First submitted 2010-04-13; First posted 2010-04-16 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Morbid Obesity
Keywords: Gastric band; Questionnaire; Post operative management; Adjustment
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gastric Band Patients
  Interventions: Behavioral: VEW Questionnaire

INTERVENTIONS:
Behavioral: VEW Questionnaire — Patient Self reported questionnaire filled in.
  Other Names: NEWLS Questionnaire

SUMMARY:
1. Background / Scientific Rationale

The VEW (Vomiting, Eating, and Weight Loss) Questionnaire has been developed as a method for the assessment of post bariatric surgery patients, as well as a research tool into the eating behaviour of these patients.

Objective VEW Questionnaire Premise If used optimally the VEW score is a valuable tool for patients who have had Laparoscopic Gastric Band Surgery (LAGB). The VEW score will be able to assist clinicians treating patients with a LAGB, specifically the Swedish Adjustable Gastric Band (SAGB), by providing them a tool to enhance patient outcomes. By using the information gained from the VEW questionnaire we can assess many areas of the eating behavior, and adjustment outcomes in patients with Gastric Bands.

Hypotheses:

* The VEW questionnaire aids in the assessment of the need for gastric band adjustment (up or down in volume)

  * Comparison of patient factors in those who have had a

    1. good outcome (increased weight loss)
    2. bad outcomes (vomiting, low weight loss, maladaption), from a gastric band fluid addition
  * In patients who have had a bad outcome, which factors are more predictive?
* Fewer Complications associated with Gastric Band Adjustments

  * Obstruction
  * Need for urgent deflation
  * Pain on eating
  * Lowering incidence of inappropriate fills
  * Lower incidence of maladaption
* Eating behavior can predict long term outcomes

  o By comparison of factors in the different quartiles of weight loss (particularly top 25% cf. bottom 25%)
* Maintenance of weight loss after 12 months is best achieved by use of behavior modification via improved food tolerances and better eating behavior than by increasing restriction of the band by further adjustments. 12 months is chosen as an arbitrary time where the majority of expected weight loss (45% of expected 50-55% 0f EWL) has been achieved. It is also a time frame by which patients have learnt to use the band appropriately, and the gastric band has had time to be adjusted into its optimal range.
* The VEW questionnaire can help predict poor outcomes from a SAGB adjustment.

  * By analyzing the factors in patients who have returned both acutely (days) or at subsequent visits (weeks) and had fluid removed from their bands. These factors would include pain, vomiting, length of meals, maladaption score, fluid added, etc.

DETAILED DESCRIPTION:
1. Background / Scientific Rationale

The VEW (Vomiting, Eating, and Weight Loss) Questionnaire has been developed as a method for the assessment of post bariatric surgery patients, as well as a research tool into the eating behaviour of these patients.

Objective VEW Questionnaire Premise If used optimally the VEW score is a valuable tool for patients who have had Laparoscopic Gastric Band Surgery (LAGB). The VEW score will be able to assist clinicians treating patients with a LAGB, specifically the Swedish Adjustable Gastric Band (SAGB), by providing them a tool to enhance patient outcomes. By using the information gained from the VEW questionnaire we can assess many areas of the eating behavior, and adjustment outcomes in patients with Gastric Bands.

Hypotheses:

* The VEW questionnaire aids in the assessment of the need for gastric band adjustment (up or down in volume)

  o Comparison of patient factors in those who have had a
  1. good outcome (increased weight loss)
  2. bad outcomes (vomiting, low weight loss, maladaption), from a gastric band fluid addition o In patients who have had a bad outcome, which factors are more predictive?
* Fewer Complications associated with Gastric Band Adjustments o Obstruction o Need for urgent deflation

  o Pain on eating
  * Lowering incidence of inappropriate fills
  * Lower incidence of maladaption
* Eating behavior can predict long term outcomes

  * By comparison of factors in the different quartiles of weight loss (particularly top 25% cf. bottom 25%)
* Maintenance of weight loss after 12 months is best achieved by use of behavior modification via improved food tolerances and better eating behavior than by increasing restriction of the band by further adjustments. 12 months is chosen as an arbitrary time where the majority of expected weight loss (45% of expected 50-55% 0f EWL) has been achieved. It is also a time frame by which patients have learnt to use the band appropriately, and the gastric band has had time to be adjusted into its optimal range.
* The VEW questionnaire can help predict poor outcomes from a SAGB adjustment.

  * By analyzing the factors in patients who have returned both acutely (days) or at subsequent visits (weeks) and had fluid removed from their bands. These factors would include pain, vomiting, length of meals, maladaption score, fluid added, etc.

    3. Study Population, including Inclusion/Exclusion There are 507 patients that are eligible for inclusion to this study. The patients that will be included are only those patients that are eligible for a LAGB adjustment (thus excluding preoperative and the first post-operative visit) and have presented for review by the treating surgeon (single surgeon) in the year 2009. All non-gastric band and non-SAGB gastric bands have been excluded. Assessments by dietitians and psychologists have also been excluded.

    4. Study Procedures Initial Patient consent for the VEW questionnaire is obtained in consultation with the treating surgeon and dietician where the expectation, benefits and knowledge are explained and confirmed. This occurs prior to the need for adjustments, that is, during the preoperative period. To date there have been no patients that have not participated with the questionnaire.

The VEW questionnaire is handed out to all eligible (please see description for eligibility in point three) upon arrival to the clinic. Patients are given five minutes to fill out the questionnaire which is then brought into the consultation with them.

Patient care and treatment is done with the strictest adherence to the Declaration of Helsinki and in the aim of developing new and better guidelines for Best Practice for the treatment of patients who have had a LAGB.

5. Duration of Study Twelve months starting 1st January 2009-31st December 2009.

6. Procedure Type

The VEW score study is limited to patients that have had LAGB specifically the Swedish Adjustable Gastric Band (SAGB):

o SAGB -VC

* SABG -QC
* SAGB - 2100 The VEW questionnaire is used following all bariatric procedures but the study would be limited to the above subset of patients.

  7. Primary / Secondary Safety and Efficacy Endpoints

Primary Efficacy Endpoints:

* Optimal gastric band adjustment tailored for the patient for no pain on eating, no obstructions and urgent deflation of the band
* Inappropriate adjustment of the LAGB
* Identify and Decrease the incidence of maladaptive eating behaviours

Secondary Efficacy Endpoints:

* Excess Weight loss at 3, 6, 12 months
* Eating behaviour at 3,6,12 months
* Incidence of Vomiting
* Fill frequency and outcome

  8. Statistical Analysis Plan

Due to the significant amount of data that is currently contained in the North Eastern Weightloss Surgery database I have decided to narrow the parameters to the following for this particular study:

o All patients will be broken into two arms, one control arm and one trial arm.

o The outcomes that will be looked for are:

1. Number of adjustments per patient
2. Efficacy of the adjustments
3. Excess Weight Loss (EWL)
4. Eating behaviour and its changes
5. Food tolerances (as per the Moore-Bohn Food tolerance scale)

9. Safety Considerations and Reporting There are no safety considerations relating tho the use of the VEW questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received a Swedish Adjustable Gastric gastric band

Exclusion Criteria:

* Patients who haven't received a Swedish Adjustable Gastric Band

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have received a Swedish Adjustable Gastric band at North Eastern Weight Loss Surgery
Sampling Method: Probability Sample
Enrollment: 361 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 1 year

SECONDARY OUTCOMES:
Vomiting Frequency | 12 months
Maladaptive eating | 12 months
  Evaluation of any change in dietary habits
Gastric Band adjustments | 12 months
  Number of adjustments

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Moore, MBBS FRACS, Principal Investigator — North Eastern Weight Loss Surgery
Locations (1):
- North Eastern Weight Loss Surgery, Melbourne, Victoria, Australia